CLINICAL TRIAL: NCT01548625
Title: Cardiovascular Effects of Incremental Diesel Exhaust Inhalation in Middle-Aged Healthy GSTM1 Null Human Volunteers
Status: Completed | Type: Observational
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Haiyan Tong, Principal Investigator, Environmental Protection Agency (EPA)
Other Study IDs: DE pilot
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2012-03

CONDITIONS: Healthy
Keywords: risk of cardiovascular events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy middle-aged human volunteers

SUMMARY:
Purpose: A growing body of epidemiological data suggests an increased risk of cardiovascular events associated with air pollutants. Reactive oxygen species (ROS) have been implicated as a potential mechanism for the adverse effects of air pollutants and genetic polymorphisms of the glutathione-s-transferases (GSTs) have been shown to participate in the antioxidant defenses to air pollutants. This study examined the dose effects of diesel exhaust exposure on the cardiovascular system in healthy middle-aged subjects.

Participants: Six healthy 50-75 year-old male and female subjects with GSTM1 null genotype had 3 sequential exposures to the diesel exhausts at concentrations approximately 100 µg/m3, 200 µg/m3, and 300 µg/m3 for 2 hours with a about 2 weeks of interval between exposures.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old generally healthy male and female.
* Normal resting ECG.
* Oxygen saturation greater than 94% at the time of physical exam.

Exclusion Criteria:

* A history of angina, cardiac arrhythmias, and ischemic myocardial infarction or coronary bypass surgery.
* Cardiac pacemaker.
* Uncontrolled hypertension (> 150 systolic, > 90 diastolic).
* Neurodegenerative diseases such as Parkinson's and Alzheimer disease.
* A history of chronic illnesses such as diabetes, cancer, rheumatologic diseases, immunodeficiency state, known cardiovascular disease, chronic respiratory diseases such as chronic obstructive pulmonary disease or severe asthma.
* History of bleeding diathesis.
* Currently taking HMG-CoA reductase inhibitors for hyperlipidemia including lovastatin, pravastatin, simvastatin, and atorvastatin.
* Currently taking beta-blockers to control hypertension and/or arrhythmias.
* Use of oral anticoagulants.
* Participants must refrain from all over-the-counter NSAIDs for a period of two weeks prior to exposure. Low-dose aspirin will be acceptable. Medications not specifically mentioned here may be reviewed by the investigators prior to a participant's inclusion in the study.
* Subjects who are currently smoking or have smoking history within 1 year of study (defined as more than one pack of cigarettes in the past year).
* Subject is pregnant, attempting to become pregnant or breastfeeding.
* No exposure will be conducted within 4 weeks of a respiratory tract infection.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy 50-75 year-old male and female subjects with GSTM1 null genotype.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Vascular effects of DE exposure | One hour before and 1 hour after DE exposure
  Brachial artery ultrasound was performed to measure vascular effects of DE exposure

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States